CLINICAL TRIAL: NCT05440643
Title: A Phase I/II Trial in 3 Parts Assessing the Safety, Tolerability, and Efficacy of a Once-daily Peanut Sublingual Immunotherapy (SLIT) Tablet in Adults, Adolescents, and Children With Peanut Allergy
Brief Title: Peanut Sublingual Immunotherapy (SLIT)-Tablet for Treatment of Peanut Allergy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT-01
Record Dates: First submitted 2022-06-17; First posted 2022-07-01 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Peanut Allergy
Keywords: Peanut allergy; Children; Adolescent; Adult
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Part 1 and 2 is sequential Part 3 is parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 and 2 is open label. Part 3 is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1: Cohort 1 (Experimental): Adults and adolescents - peanut SLIT-tablet once daily for 2 weeks
  Interventions: Biological: Peanut SLIT-tablet
- Part 1: Cohort 2 (Experimental): Adults and adolescents - peanut SLIT-tablet once daily for 2 weeks
  Interventions: Biological: Peanut SLIT-tablet
- Part 1: Cohort 3 (Experimental): Adults and adolescents - peanut SLIT-tablet once daily for 2 weeks
  Interventions: Biological: Peanut SLIT-tablet
- Part 1: Cohort 4 (Experimental): Adults and adolescents - peanut SLIT-tablet once daily for 2 weeks
  Interventions: Biological: Peanut SLIT-tablet
- Part 1: Cohort 5 (Experimental): Adults and adolescents - peanut SLIT-tablet once daily for 2 weeks
  Interventions: Biological: Peanut SLIT-tablet
- Part 2: Cohort 6 (Experimental): Adults - UDR with once daily peanut SLIT-tablet
  Interventions: Biological: Peanut SLIT-tablet
- Part 2: Cohort 7 (Experimental): Adolescents - UDR with once daily peanut SLIT-tablet
  Interventions: Biological: Peanut SLIT-tablet
- Part 2: Cohort 8 (Experimental): Children - UDR with once daily peanut SLIT-tablet
  Interventions: Biological: Peanut SLIT-tablet
- Part 2: Cohort 9 (Experimental): Highly sensitized Adults/Adolescents - UDR with once daily peanut SLIT-tablet
  Interventions: Biological: Peanut SLIT-tablet
- Part 2: Cohort 10 (Experimental): Highly sensitized Children - UDR with once daily peanut SLIT-tablet
  Interventions: Biological: Peanut SLIT-tablet
- Part 3: Maintenance A (Experimental): UDR A + maintenance dose A
  Interventions: Biological: Peanut SLIT-tablet
- Part 3: Maintenance B (Experimental): UDR B + maintenance dose B
  Interventions: Biological: Peanut SLIT-tablet
- Part 3: Placebo (Placebo Comparator): Placebo UDR + placebo maintenance
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Peanut SLIT-tablet — Peanut extract
  Arms: Part 1: Cohort 1; Part 1: Cohort 2; Part 1: Cohort 3; Part 1: Cohort 4; Part 1: Cohort 5; Part 2: Cohort 10; Part 2: Cohort 6; Part 2: Cohort 7; Part 2: Cohort 8; Part 2: Cohort 9; Part 3: Maintenance A; Part 3: Maintenance B
Other: Placebo — Placebo
  Arms: Part 3: Placebo

SUMMARY:
This clinical research study investigates the safety, tolerability and efficacy of a peanut SLIT-tablet in adults, adolescents, and children with peanut allergy.

DETAILED DESCRIPTION:
This is a phase I/II, dose-escalation, multi-site trial including subjects with peanut allergy confirmed by screening double-blind, placebo-controlled food challenge. The trial is conducted in 3 parts; part 1 will determine the entry dose of the up-dosing regimen (UDR) in adults and adolescents; part 2 will characterize the tolerability of the up-dosing regimen in adults, adolescents and children; part 3 will evaluate the efficacy of 2 maintenance doses of the SLIT-tablet primarily in adolescents and children; a small number of adults may also be included.

Peanut SLIT tablets administered as 9 doses covering a 4000-fold increase in dose will be used in the study.

In part 1, subjects will receive a peanut SLIT-tablet with one of five doses once daily for 2 weeks.

In part 2, subjects will receive a series of increasing doses of the peanut SLIT-tablet, where each dose is taken once daily for 2 weeks. The entry dose for the up-dosing regimen will be determined from part 1.

In part 3, subjects will be randomized into 3 treatment groups (UDR and Maintenance A, UDR and Maintenance B, Placebo UDR and Placebo). Subjects will receive a series of increasing doses of the peanut SLIT-tablet , where each dose is taken once daily for 2 weeks, followed by Maintenance A or B once daily for 24 weeks; or the corresponding Placebo.

The trial will consist of up to 10 cohorts (part 1 is cohort 1-5; part 2 is cohort 6-10) and 3 treatment groups in part 3.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

Subjects are eligible to be included in the trial only if all the following criteria apply:

* Part 1: Male or female aged 12 through 65 years (inclusive) on the day of enrollment Part 2: Male or female aged 4 through 65 years (inclusive) on the day of enrollment Part 3: Male or female aged 4 through 65 years (inclusive) on the day of randomization
* Documented clinical history of an IgE-mediated allergic reaction towards peanut- containing food
* Peanut-specific serum IgE ≥ 0.7 kU/L at screening measured at central laboratory
* Skin prick test to peanut ≥ 5 mm at screening
* Cohorts 1-8: Experience dose-limiting symptoms at the 10 mg, 30 mg or 100 mg challenge dose of peanut protein on screening DBPCFC Cohorts 9-10: Experience dose-limiting symptoms at the 1 mg or 3 mg challenge dose of peanut protein on the screening DBPCFC Part 3: Experience dose-limiting symptoms at the 3 mg, 10 mg, 30 mg or 100 mg challenge dose of peanut protein on screening DBPCFC

KEY EXCLUSION CRITERIA:

Subjects are excluded from the trial if any of the following criteria apply:

* Diagnosis or history of eosinophilic esophagitis
* Uncontrolled asthma as defined by the Asthma Control Test questionnaire with a score of 19 or below at enrollment (subjects with a diagnosis of asthma only)
* All subjects ≥ 5 years old with FEV1 or PEFR < 70% of predicted value at enrollment Subjects 4 years old with a history of recurrent wheeze requiring inhaled corticosteroids for 2 consecutive weeks or more within 3 months prior to enrollment
* Up-dosing with any allergy immunotherapy product. Maintenance dose of any subcutaneous immunotherapy product other than peanut is allowed
* History of peanut oral immunotherapy within the last 12 months prior to visit 1
* Chronic or acute oral inflammation at enrollment
* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* Currently using any prohibited medication on the list of prohibited medication
* Part 1 and 2: Allergic symptoms in reaction to the placebo part of the screening DBPCFC Part 3: Dose-limiting allergic symptoms in reaction to the placebo part of the screening DBPCFC
* History of severe or life-threatening episode of anaphylaxis or anaphylactic shock within 60 days of the screening DBPCFC
* Part 1 and 2: Asthma according to below criteria:

  * Severe asthma as per the current GINA guidelines
  * Uncontrolled or poorly controlled asthma as per the current GINA guidelines
  * Asthma that requires more than a daily dose above 800 µg of inhaled budesonide (or clinically comparable inhaled corticosteroids)
  * History of 2 or more systemic corticosteroid courses within 6 months of screening
  * Prior intubation/mechanical ventilation for asthma
  * Emergency room visit or hospitalization for asthma in the 12 months prior to screening
  * Any history of a life-threatening asthma attack
* Part 3: Asthma fulfilling the below criteria:

  * History of 2 or more systemic corticosteroid courses within 6 months of screening
  * Prior intubation/mechanical ventilation for asthma
  * Emergency room visit or hospitalization for asthma in the 12 months prior to screening
  * Any history of a life-threatening asthma attack
  * (US only) Severe asthma as per the current GINA guidelines
  * (US only) Uncontrolled or poorly controlled asthma as per the current GINA guidelines
  * (US only) Asthma that requires more than a daily maintenance dose above 800 μg of inhaled budesonide (or clinically comparable inhaled corticosteroids)

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Dose tolerability response rate | 2 weeks per dose
  The dose tolerability response rate is defined as the percentage of subjects who experience at most moderate local application site reactions after the last peanut SLIT-tablet intake of the dose step. Local application site reactions are treatment-related adverse events occurring in close proximity to the application site of the SLIT-tablet with a temporal relationship to tablet administration.
Part 3: TD-600 response rate | After 24 weeks of maintenance treatment, up to 48 weeks.
  The TD (tolerated dose)-600 response rate is defined as the percentage of subjects able to consume 600 mg (1044 mg cumulative) peanut protein without dose-limiting symptoms at the exit double-blind placebo-controlled food challenge (DBPCFC) after 24 weeks of maintenance treatment. Subjects that do not complete the exit DBPCFC are classified as non-responders.

SECONDARY OUTCOMES:
Part 1, 2 and 3: Treatment-emergent adverse events | Part 1 and 2: 2 weeks per dose; Part 3: from first IMP intake to 7 days after last IMP intake, up to 48 weeks.
  An adverse event is any untoward medical occurrence in a clinical trial subject and which does not necessarily have a causal relationship with the administered investigational medicinal product (IMP). A treatment-emergent adverse event has a start date on or after the time of first IMP intake and no later than 7 days after the last IMP intake.
Part 3: TD-300 response rate | After 24 weeks of maintenance treatment, up to 48 weeks.
  The TD-300 response rate is defined as the percentage of subjects able to consume 300 mg (444 mg cumulative) peanut protein without dose-limiting symptoms at the exit DBPCFC after 24 weeks of maintenance treatment. Subjects that do not complete the exit DBPCFC are classified as non-responders.
Part 3: TD-1000 response rate | After 24 weeks of maintenance treatment, up to 48 weeks.
  The TD-1000 response rate is defined as the percentage of subjects able to consume 1000 mg (2044 mg cumulative) peanut protein without dose-limiting symptoms at the exit DBPCFC after 24 weeks of maintenance treatment. Subjects that do not complete the exit DBPCFC are classified as non-responders.
Part 3: TD-2000 response rate | After 24 weeks of maintenance treatment, up to 48 weeks.
  The TD-2000 response rate is defined as the percentage of subjects able to consume 2000 mg (4044 mg cumulative) peanut protein without dose-limiting symptoms at the exit DBPCFC after 24 weeks of maintenance treatment. Subjects that do not complete the exit DBPCFC are classified as non-responders.
Part 3: Maximum tolerated dose of peanut protein during DBPCFC | At screening, 1 - 3 weeks, and after 24 weeks of maintenance treatment, up to 48 weeks.
  The highest single challenge dose of peanut protein that a subject can consume without experiencing dose-limiting symptoms during the DBPCFC.
Part 3: Maximum severity of symptoms at each challenge dose of peanut protein during DBPCFC | At screening, 1 - 3 weeks, and after 24 weeks of maintenance treatment, up to 48 weeks.
  The highest severity of any symptom experienced at any challenge dose during the DBPCFC. Possible values are 0=none, 1=mild, 2=moderate or 3=severe.
Part 3: Response rate - use of epinephrine as rescue medication during exit DBPCFC | After 24 weeks of maintenance treatment, up to 48 weeks.
  The response rate is defined as the percentage of subjects that receive epinephrine as rescue medication during the exit DBPCFC.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Kim, MD, Principal Investigator — University of North Carolina
Locations (40):
- United States (31):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles - USC School of Medicine, Los Angeles, California
  - UCLA - Pediatrics, Los Angeles, California
  - Stanford University - Lucile Packard Children's Hospital, Palo Alto, California
  - Peninsula Research Associates (PRA), Rolling Hills Estates, California
  - Eastern Virginia Medical School - Children's Hospital, San Diego, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Quality Research of South Florida, Hialeah, Florida
  - MOORE-PH Dermatology - Clinical Research, Tampa, Florida
  - USF Asthma Allergy and Immunology Clinical Research Unit, Tampa, Florida
  - Center for Advance Pediatrics, Atlanta, Georgia
  - Ann Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - Family Allergy Asthma Research Institute, Louisville, Kentucky
  - Velocity Clinical Research - Lafayette, Lafayette, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Asthma, Allergy and Sinus Center, White Marsh, Maryland
  - Boston Food Allergy Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Northwell Health, Great Neck, New York
  - NYU Langone Health - Fink Children's Ambulatory Care Center, New York, New York
  - Icahn School of Medicine at Mt. Sinai, Pediatric Allergy, Kravis Children Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Aventiv research, Inc, Columbus, Ohio
  - Children's Hospital of Philadephia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburg of UPMC - Immunology and Rheumatology, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Baylor College of Medicine (BCM) Texas Children's Hospital Pediatrics and Immunology, Houston, Texas
- Canada (9):
  - BC Children's Hospital, Vancouver, British Colombia
  - The Children's Hospital Foundation of Manitoba, Winnipeg, Manitoba
  - Halton Pediatric Allergy, Burlington, Ontario
  - Hamilton Allergy, Hamilton, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Toronto, Ontario
  - McGill University Health Centre (MUHC) - Research Institute (RI-MUHC), Montreal, Quebec
  - CHU-Saint-Justine, Montreal, Quebec
  - Clinique Specialisee en Allergie de la Capitale, Québec